CLINICAL TRIAL: NCT03224130
Title: Supplement to Hospital to Home Outcomes (H2O): A Study to Improve the Fluidity of Transitions Between Hospital and Home
Brief Title: Supplement to Hospital to Home Outcomes
Acronym: Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H2O Supplement
Record Dates: First submitted 2016-05-10; First posted 2017-07-21 (Actual); Results first posted 2019-03-29 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Hospitalized Patients
Keywords: transitions of care; reutilization; nurse phone call
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nurse Phone Call (Experimental): Families in this arm will receive a phone call within 96 hours of discharge
  Interventions: Other: Nurse Phone Call
- Standard of Care (Active Comparator): This arm will receive standard of care.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Nurse Phone Call — We will complete a single center, parallel, randomized, standard-of-care-controlled prospective study to determine the efficacy of a one-time nurse phone call, an intervention adapted from those studied in other populations (i.e., adults, high-risk infants), in improving pediatric patient transitions from hospital to home
  Arms: Nurse Phone Call
Other: Standard of Care — Control patients will be randomized to receive standard-of-care at discharge. This care at our institution includes pediatric hospitalist to PCP (primary care physician) verbal and written communication prior to discharge, written documentation for the family regarding prescribed medication regimen, recommended follow-up with outpatient PCP and relevant consultant(s), and delivery of prescribed medications from the hospital pharmacy to the patient's bedside.
  Arms: Standard of Care

SUMMARY:
Post-discharge nurse phone call

DETAILED DESCRIPTION:
Previous work has identified barriers to successful transitions that are most meaningful to patients and families. Investigators used these learnings to iteratively adapt an existing nurse home visit program to address these barriers, and have been studying the effectiveness of the redesigned nurse home visit in a randomized control trial (NCT02081846).

ELIGIBILITY:
Inclusion Criteria:

* Patient is under 18 years of age
* Patient is admitted to Cincinnati Children's Hospital Medical Center to hospital medicine, ,community pediatrics, or adolescent medicine.

Exclusion Criteria:

* Patient to be discharged someplace other than home (e.g., residential facility, psychiatric facility)
* Patient's home residence is outside the home nursing service area
* Patient is eligible for "traditional" home nursing services
* Caregiver is non-English speaking

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 966 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Shah, MD, MSCE, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Sauers-Ford HS, Simmons JM, Shah SS; H2O Study Team. Strategies to engage stakeholders in research to improve acute care delivery. J Hosp Med. 2016 Feb;11(2):123-5. doi: 10.1002/jhm.2492. Epub 2015 Sep 28. PMID 26416164
- [Background] Tubbs-Cooley HL, Pickler RH, Simmons JM, Auger KA, Beck AF, Sauers-Ford HS, Sucharew H, Solan LG, White CM, Sherman SN, Statile AM, Shah SS; H2O Study Group. Testing a post-discharge nurse-led transitional home visit in acute care pediatrics: the Hospital-To-Home Outcomes (H2O) study protocol. J Adv Nurs. 2016 Apr;72(4):915-25. doi: 10.1111/jan.12882. Epub 2016 Jan 28. PMID 26817441
- [Background] Solan LG, Beck AF, Brunswick SA, Sauers HS, Wade-Murphy S, Simmons JM, Shah SS, Sherman SN; H2O Study Group. The Family Perspective on Hospital to Home Transitions: A Qualitative Study. Pediatrics. 2015 Dec;136(6):e1539-49. doi: 10.1542/peds.2015-2098. PMID 26620060
- [Background] Beck AF, Solan LG, Brunswick SA, Sauers-Ford H, Simmons JM, Shah S, Gold J, Sherman SN; H2O Study Group. Socioeconomic status influences the toll paediatric hospitalisations take on families: a qualitative study. BMJ Qual Saf. 2017 Apr;26(4):304-311. doi: 10.1136/bmjqs-2016-005421. Epub 2016 Jul 28. PMID 27471042
- [Background] Pickler R, Wade-Murphy S, Gold J, Tubbs-Cooley H, White CM, Statile A, Hoying C, Sauers-Ford H, Shah SS, Simmons J; H2O Study Group. A Nurse Transitional Home Visit Following Pediatric Hospitalizations. J Nurs Adm. 2016 Dec;46(12):642-647. doi: 10.1097/NNA.0000000000000420. PMID 27851705
- [Background] Sauers-Ford HS, Tubbs-Cooley H, Statile AM, Pickler RH, White CM, Wade-Murphy S, Gold JM, Shah SS, Simmons JM, Auger KA, Bachus J, Beck AF, Borell ML, Brunswick SA, Chang L, Heilman JA, Jabour JA, Khoury JC, Moore MJ, Sherman SN, Solan LG, Sucharew HJ, Sullivan KP. Optimizing a Nurse-led Transitional Home Visit Program in Preparation for a Randomized Control Trial. Pediatr Qual Saf. 2017 Jan 25;2(1):e012. doi: 10.1097/pq9.0000000000000012. eCollection 2017 Jan-Feb. PMID 30229150
- [Background] Sauers-Ford HS, Gold JM, Statile AM, Tubbs-Cooley HL, Simmons JM, Shah SS, Bell K, Pfefferman C, Moore MJ, Auger KA; H2O Study Group. Improving Recruitment and Retention Rates in a Randomized Controlled Trial. Pediatrics. 2017 May;139(5):e20162770. doi: 10.1542/peds.2016-2770. PMID 28557728
- [Background] Solan LG, Beck AF, Shardo SA, Sauers-Ford HS, Simmons JM, Shah SS, Sherman SN; H2O Study Group. Caregiver Perspectives on Communication During Hospitalization at an Academic Pediatric Institution: A Qualitative Study. J Hosp Med. 2018 May;13(5):304-310. doi: 10.12788/jhm.2919. PMID 29345256
- [Background] Shah AN, Beck AF, Sucharew HJ, Litman S, Pfefferman C, Haney J, Shah SS, Simmons JM, Auger KA; H2O Study Group. Parental Adverse Childhood Experiences and Resilience on Coping After Discharge. Pediatrics. 2018 Apr;141(4):e20172127. doi: 10.1542/peds.2017-2127. PMID 29563237
- [Background] Auger KA, Simmons JM, Tubbs-Cooley HL, Sucharew HJ, Statile AM, Pickler RH, Sauers-Ford HS, Gold JM, Khoury JC, Beck AF, Wade-Murphy S, Kuhnell P, Shah SS; H2O Trial study group. Postdischarge Nurse Home Visits and Reuse: The Hospital to Home Outcomes (H2O) Trial. Pediatrics. 2018 Jul;142(1):e20173919. doi: 10.1542/peds.2017-3919. PMID 29934295
- [Background] Auger KA, Shah SS, Tubbs-Cooley HL, Sucharew HJ, Gold JM, Wade-Murphy S, Statile AM, Bell KD, Khoury JC, Mangeot C, Simmons JM; Hospital-to-Home Outcomes Trial Study Group. Effects of a 1-Time Nurse-Led Telephone Call After Pediatric Discharge: The H2O II Randomized Clinical Trial. JAMA Pediatr. 2018 Sep 1;172(9):e181482. doi: 10.1001/jamapediatrics.2018.1482. Epub 2018 Sep 4. PMID 30039161
- [Background] Chang LV, Shah AN, Hoefgen ER, Auger KA, Weng H, Simmons JM, Shah SS, Beck AF; H2O Study Group. Lost Earnings and Nonmedical Expenses of Pediatric Hospitalizations. Pediatrics. 2018 Sep;142(3):e20180195. doi: 10.1542/peds.2018-0195. Epub 2018 Aug 13. PMID 30104421
- [Derived] Auger KA, Sucharew HJ, Simmons JM, Shah SS, Kahn RS, Beck AF; H2O Trial Study Group. Differential Impact of Home Nurse Contact After Discharge by Financial Strain, Primary Care Access, and Medical Complexity. Hosp Pediatr. 2021 Aug;11(8):791-800. doi: 10.1542/hpeds.2020-004267. PMID 34330881

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nurse Phone Call | Standard of Care
Started | 483 | 483
Completed | 483 | 482
Not Completed | 0 | 1
Not completed — consent issue | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nurse Phone Call | Standard of Care | Total
Number analyzed (Participants) | 483 | 482 | 965
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 2.4 [0.5 to 7.8] | 2.4 [0.5 to 7.8] | 2.4 [0.5 to 7.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 246 | 214 | 460
  Male | 237 | 268 | 505
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 20 | 33
  Not Hispanic or Latino | 470 | 461 | 931
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 309 | 311 | 620
  Race: Black or African American | 117 | 102 | 219
  Race: American Indian or Alaska Native | 0 | 1 | 1
  Race: Asian/Oriental or Pacific Islander | 8 | 6 | 14
  Race: Other | 49 | 61 | 110
  Race: Unknown/missing | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 483 | 482 | 965
Length of Stay [Median (Inter-Quartile Range); unit: days] — Length of hospital stay in days.
  days | 2 [1 to 2] | 2 [1 to 2] | 2 [1 to 2]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Occurrence of Unplanned Re-hospitalization and/or Any Emergency/Urgent Care Visits Within 30 Days of Hospital Discharge
Description: The dependent variable will be a dichotomized indicator of any occurrence of unplanned rehospitalization, ED or urgent care visit within 30-days post-discharge (i.e. unplanned reutilization). Differences in this outcome between intervention and control groups will be evaluated using logistic regression with the stratification variables (neighborhood poverty and state)
Time Frame: 30 days post-discharge
Population: The analysis population includes the total 966 (483 intervention, 483 control) randomized excluding the one subject withdrawn in the control group after randomization due to invalid consent at 14-day follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Nurse Phone Call | Standard of Care
Number analyzed (Participants) | 483 | 482
Participants | 77 | 63
Statistical Analysis 1: Comparison: Nurse Phone Call vs Standard of Care; Test type: Superiority; p = 0.21, Regression, Logistic

2. Secondary Outcome: Post-Discharge Coping Scale
Description: Post-Discharge Difficulty Coping Scale (Weiss, et. al): measured at 14 day post-discharge phone call. Post-Discharge Coping Difficulty Scale uses an 11 point scaling format (0-10) with total scores ranging from 0 to 100. Higher scores represent greater coping difficulty. Differences between intervention and control groups on this outcome at 14-day post-discharge are evaluated using a linear regression model with the stratification variables (census tract poverty and state of residence).
Time Frame: 14 days post-discharge
Population: The analysis population includes the total subjects completing the 14-day phone call survey for this outcome. Of the total randomized (966: 483 intervention, 483 control), 26 were excluded from the intervention group and 23 from the control group.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Nurse Phone Call | Standard of Care
Number analyzed (Participants) | 457 | 460
units on a scale | 14.3 [12.8 to 15.8] | 15.2 [13.7 to 16.7]
Statistical Analysis 1: Comparison: Nurse Phone Call vs Standard of Care; Test type: Superiority; p = 0.31, Regression, Linear

3. Secondary Outcome: Number of Days Until Normalcy
Description: Number of days until normalcy: measured at post discharge phone call. Parents asked to recall the number of days it took to "return to a 'normal' routine" including the return to work and school (with option of not yet be back to normal).
Time Frame: 14 days post-discharge
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: days
Arm/Group | Nurse Phone Call | Standard of Care
Number analyzed (Participants) | 457 | 460
days | 3.9 [3.5 to 4.2] | 4.2 [3.8 to 4.6]
Statistical Analysis 1: Comparison: Nurse Phone Call vs Standard of Care; Test type: Superiority; p = 0.24, censored Poisson model

4. Secondary Outcome: Red Flags Remembered
Description: This was measured at the 14 day post-discharge phone call survey. Parents were asked to recall "any red flags or warning signs" to indicate the "child's condition was getting worse." The number of red flags recalled could range from 0-10 depending on the template used. The template was a home visit guideline for nurses to use that was specific to the child's illness. For example, if the child had bronchiolitis the nurse would use the template "bronchiolitis/croup/pneumonia" to guide them through the visit. Higher values (i.e., the greater number of red flags remembered) represent a better outcome.
Time Frame: 14 days post-discharge
Population: The analysis population includes the total subjects completing the 14-day phone call survey for this outcome. Of the total randomized (966: 483 intervention, 483 control), 25 were excluded from the intervention group and 23 from the control group.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Nurse Phone Call | Standard of Care
Number analyzed (Participants) | 458 | 460
units on a scale | 1.8 [1.7 to 2.0] | 1.5 [1.4 to 1.6]
Statistical Analysis 1: Comparison: Nurse Phone Call vs Standard of Care; Test type: Superiority; p < 0.01, Poisson model

5. Secondary Outcome: Number of Participants With Occurrence(s) of an Unplanned Readmission Within 30 Days Post-discharge
Description: Occurrence(s) of an unplanned readmission within 30 days post-discharge.
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nurse Phone Call | Standard of Care
Number analyzed (Participants) | 483 | 482
Participants | 32 | 27
Statistical Analysis 1: Comparison: Nurse Phone Call vs Standard of Care; Test type: Superiority; p = 0.50, Regression, Logistic

6. Secondary Outcome: Number of Participants With Occurrence(s) of an Emergency Department Visit Within 30 Days Post-discharge
Description: Occurence(s) of an ED visit within 30 days post-discharge
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nurse Phone Call | Standard of Care
Number analyzed (Participants) | 483 | 482
Participants | 35 | 35
Statistical Analysis 1: Comparison: Nurse Phone Call vs Standard of Care; Test type: Superiority; p = 0.998, Regression, Logistic

7. Secondary Outcome: Number of Participants With Occurrence(s) of 14-day Unplanned Healthcare Utilization
Description: Occurrence(s) of 14-day unplanned healthcare utilization defined by unplanned re-hospitalization and/or any emergency/urgent care visit within 14 days or parent report of an unplanned visit to one of these places. Parent report is collected at the 14 day follow-up phone call.
Time Frame: 14 days post-discharge
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nurse Phone Call | Standard of Care
Number analyzed (Participants) | 483 | 482
Participants | 71 | 72
Statistical Analysis 1: Comparison: Nurse Phone Call vs Standard of Care; Test type: Superiority; p = 0.92, Regression, Logistic

ADVERSE EVENTS:
Time Frame: enrollment to 30 days post discharge
Description: As this study involved minimal risk to the individuals recruited, we relied solely on caregiver report of any adverse event or serious adverse event during the study encounter (enrollment to 30 days post discharge). All-Cause Mortality was not monitored/assessed.
Arm/Group | Nurse Phone Call | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/483 | 0/483
Other Adverse Events (participants affected / at risk) | 0/483 | 0/483

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT03224130/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT03224130/SAP_001.pdf